CLINICAL TRIAL: NCT06870981
Title: Improving Growth and Neurodevelopment of Very Low Birth Weight Infants Through Precision Nutrition: The Optimizing Nutrition and Milk (Opti-NuM) Project
Brief Title: Optimizing Nutrition and Milk (Opti-NuM) Project
Acronym: Opti-NuM
Status: Recruiting | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Mount Sinai Hospital, Canada (Other); Sunnybrook Health Sciences Centre (Other); University of Toronto (Other); University of Manitoba (Other); Stanford University (Other); University of California, San Diego (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Deborah O'Connor, Senior Associate Scientist, The Hospital for Sick Children
Other Study IDs: 4842; 5R01HD111018-03 (NIH)
Record Dates: First submitted 2025-02-03; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Very Low Birth Weight Baby; Early Nutrition and the Preterm Infant; Nutritional Requirements; Human Milk Fortification; Human Milk Microbiome; Human Milk Feeding; Human Milk Nutrition; Growth &Amp; Development
Keywords: Very Low Birth Weight Infants; Early nutrition and the preterm infant; Human milk feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — 1. Human milk
  2. Stool
  3. Residual plasma
  4. Buccal cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants of the MaxiMoM Platform Trials: Secondary data use and biospecimens from participants of the MaxiMoM Platform Trials are infants born 1500g or less (infant weight), born in the Greater Toronto Area.
  Interventions: Other: Opti-NuM is an observational secondary use of data/samples study, the investigators will analyze information and specimens from the MaxiMoM platform RCTs. No interventions form part of this study.

INTERVENTIONS:
Other: Opti-NuM is an observational secondary use of data/samples study, the investigators will analyze information and specimens from the MaxiMoM platform RCTs. No interventions form part of this study.

SUMMARY:
Early nutrition critically influences growth, neurodevelopment and morbidity among infants born of very low birth weight (VLBW), but current one-size-fits-all feeding regimes do not optimally support these vulnerable infants. There is increasing interest in "precision nutrition" approaches, but it is unclear which Human Milk (HM) components require personalized adjustment of doses. Previous efforts have focused on macronutrients, but HM also contains essential micronutrients as well as non-nutrient bioactive components that shape the gut microbiome. Further, it is unclear if or how parental factors (e.g. body mass index, diet) and infant factors (e.g. genetics, gut microbiota, sex, acuity) influence relationships between early nutrition and growth, neurodevelopment and morbidity. Understanding these complex relationships is paramount to developing effective personalized HM feeding strategies for VLBW infants. This is the overarching goal of the proposed Optimizing Nutrition and Milk (Opti-NuM) Project.

The Opti-NuM Project brings together two established research platforms with complementary expertise and resources: 1) the MaxiMoM Program* with its clinically embedded translational neonatal feeding trial network in Toronto (Dr. Deborah O'Connor, Dr. Sharon Unger) and 2) the International Milk Composition (IMiC) Consortium, a world-renowned multidisciplinary network of HM researchers and data scientists collaborating to understand how the myriad of HM components contribute "as a whole" to infant growth and development, using systems biology and machine learning approaches. Members of the IMiC Corsortium that will work with on this study are located at the University of Manitoba (Dr. Meghan Azad), University of California (Dr. Lars Bode) and Stanford (Dr. Nima Aghaeepour).

DETAILED DESCRIPTION:
Observational study mode:

The Opti-NuM Project is a retrospective secondary data/sample use study.

Time perspective:

Secondary use data and biospecimens accruing from the 2 completed studies DoMINO and OptiMOM (NCT02137473) and 1 ongoing RCT MaxiMoM (NCT05308134) are included in this project.

Sampling method:

This project is a secondary use of data/samples, from a cohort consisting of participants of the MaxiMoM Platform RCTs.

ELIGIBILITY:
Inclusion Criteria:

• Secondary data and biospecimens from participants of the MaxiMoM Platform RCTs

Exclusion Criteria:

• Data and biospecimens from infants who are not enrolled in the three trials are eligible for this project.

Ages: 1 Hour to 21 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Very Low Birth Weight infants
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2010-10-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Cognitive composite score on the Bayley Scales of Infant and Toddler Development. | At 18-24 months CA
  Our primary outcome is the cognitive composite score on the Bayley Scales of Infant and Toddler Development collected from the medical record or by home-visit by our research staff. The Bayley is the most widely used instrument globally by clinicians and researchers to assess developmental functioning of infants, toddlers and young children across cognitive, language (receptive, expressive) and motor (fine, gross) domains. Cognitive, language and motor composite scores will be standardized to a mean of 100 with a standard deviation of 15.
  The range on the composite Bayle Scores is from less than 0.1 to more than 99.9 percentile. A score lower than the 10th percentile indicates developmental delay.

SECONDARY OUTCOMES:
Language composite score from the Bayley Scales of Infant and Toddler Development | At 18-24 months CA
  Language composite score from the Bayley Scales of Infant and Toddler Development. The range on the composite Bayle Scores is from less than 0.1 to more than 99.9 percentile. A score lower than the 10th percentile indicates developmental delay.
Motor composite score from the Bayley Scales of Infant and Toddler Development | At 18-24 months CA
  Motor composite score from the Bayley Scales of Infant and Toddler Development. The range on the composite Bayle Scores is from less than 0.1 to more than 99.9 percentile. A score lower than the 10th percentile indicates developmental delay.
Weight (g) | Initial hospitalization, approximately 50 days; at 4 months and 18-24 months CA clinic visit.
  Weight gains serve as early indicators of the effectiveness of early nutrition and are on the causal pathway to neurodevelopment. Daily weights are prospectively extracted from medical records.
Length (cm) | Initial hospitalization, approximately 50 days; at 4 months and 18-24 months CA clinic visit.
  Length gains serve as early indicators of the effectiveness of early nutrition and are on the causal pathway to neurodevelopment. Weekly length is determined by research staff using length boards and standardized procedures.
Head circumference (cm) | Initial hospitalization, approximately 50 days; at 4 months and 18-24 months CA clinic visit.
  Head circumference (HC) gains serve as early indicators of the effectiveness of early nutrition and are on the causal pathway to neurodevelopment. Weekly HC measurements are determined by research staff using non-stretchable tape measures and standardized procedures.
Serious morbidities | During hospital stay, an average of 60 days.
  Serious morbidities including late-onset sepsis (>day 5, positive blood or cerebrospinal fluid culture), NEC (Bell stage ≥II), chronic lung disease (respiratory support at 36 weeks) and retinopathy of prematurity requiring treatment are collected prospectively from the medical chart.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah L O'Connor, PhD, RN, Principal Investigator — The Hospital for Sick Children
Locations (6):
- United States (2):
  - Stanford University, Palo Alto, California
  - University of California - San Diego, San Diego, California
- Canada (4):
  - University of Manitoba, Winnipeg, Manitoba
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Data transfer will take place via Secure File Transfer Protocol (SFTP). Sub-agreements which cover data and sample sharing and confidentiality is in place.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: December 2024 to December 2027
Access Criteria: During the Opti-NuM project the following institutions will be involved in data and sample analysis as indicated. Data sharing will take place through SFTP, bio specimens will be shipped for analyses.
  * The Hospital for Sick Children (Lead, Deborah O'Connor PhD RD): Both data and sample analysis
  * The University of Toronto (Lead, Deborah O'Connor PhD RD): Both data and sample analysis
  * The University of Manitoba (Lead, Meghan Azad PhD): Data analysis; No sample analysis
  * Stanford University (Lead, Nima Aghaeepour PhD): Data analysis; No sample analysis
  * University of California (Lead, Lars Bode PhD): Oligosaccharide analysis of human milk samples only. No data provided to this site.

REFERENCES:
- [Background] O'Connor DL, Kiss A, Tomlinson C, Bando N, Bayliss A, Campbell DM, Daneman A, Francis J, Kotsopoulos K, Shah PS, Vaz S, Williams B, Unger S; OptiMoM Feeding Group. Nutrient enrichment of human milk with human and bovine milk-based fortifiers for infants born weighing <1250 g: a randomized clinical trial. Am J Clin Nutr. 2018 Jul 1;108(1):108-116. doi: 10.1093/ajcn/nqy067. PMID 29878061
- [Background] O'Connor DL, Gibbins S, Kiss A, Bando N, Brennan-Donnan J, Ng E, Campbell DM, Vaz S, Fusch C, Asztalos E, Church P, Kelly E, Ly L, Daneman A, Unger S; GTA DoMINO Feeding Group. Effect of Supplemental Donor Human Milk Compared With Preterm Formula on Neurodevelopment of Very Low-Birth-Weight Infants at 18 Months: A Randomized Clinical Trial. JAMA. 2016 Nov 8;316(18):1897-1905. doi: 10.1001/jama.2016.16144. PMID 27825008
- See also: MaxiMoM Research Platform — https://www.maximom-research.com/